CLINICAL TRIAL: NCT06866470
Title: Effects of Massage and Progressive Muscle Relaxation Exercise on the Severity and Frequency of Muscle Cramps in Hemodialysis Patients: A Randomized Controlled Trial
Brief Title: Muscle Cramps in Hemodialysis Patients: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: tXazkY4r
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Nursing Caries; Hemodialysis Complication; Exercise Addiction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stretching exercise group (Experimental): stretching exercise group
  Interventions: Behavioral: relaxation group

INTERVENTIONS:
Behavioral: relaxation group — exercise group

SUMMARY:
Muscle cramps are a common and distressing issue among hemodialysis patients, significantly impacting their quality of life. Non-pharmacological approaches are increasingly being explored to alleviate these symptoms. Massage therapy and progressive muscle relaxation exercises are among the interventions that may help reduce the frequency and severity of cramps by promoting muscle relaxation. However, their effectiveness in hemodialysis patients has not been sufficiently studied.

This randomized controlled trial aims to evaluate the effects of massage and progressive muscle relaxation exercises on the frequency and severity of muscle cramps in hemodialysis patients. The findings are expected to contribute to evidence-based practices in symptom management.

DETAILED DESCRIPTION:
Method Study Design and Setting This study will be conducted using a quasi-experimental design to evaluate the effects of foot massage and progressive muscle relaxation exercises (PMRE) on muscle cramps in hemodialysis patients. The study will take place at the hemodialysis center of Istanbul Gaziosmanpasa Training and Research Hospital between February and August 2025.

Population and Sample The study population consists of all hemodialysis patients registered at the study center, while the sample will include voluntary hemodialysis patients with similar demographic characteristics and dialysis treatment methods who meet the study criteria. Since no identical study exists in the literature, a power analysis was conducted to determine the sample size required to show a significant difference in the reduction of the mean number of cramps (effect size = 1), with 80% power and a 5% Type I error rate. Accordingly, 30 patients per group (massage group, PMRE group, and control group), totaling 90 patients, were planned for inclusion in the study.

Inclusion criteria:

Aged 18 years and older Receiving chronic hemodialysis treatment Experiencing muscle cramps in the last three months No physical or mental health conditions preventing communication

Exclusion criteria:

Presence of acute health issues requiring additional pharmacological treatment Inability to complete PMRE or massage applications Randomization Patients who meet the inclusion criteria and provide consent will undergo an initial interview conducted by the primary researcher, during which baseline data will be collected. Patients will be stratified based on dialysis session frequency, cramp frequency, age, and gender. To ensure homogeneity, patients will be asked about the frequency and severity of cramps experienced in the previous week. Based on the mean cramp frequency and severity scores obtained, hemodialysis patients will be categorized accordingly. Group assignments will be determined using simple randomization via an online tool (www.randomizer.org).

Data Collection Tools Demographic Information Form: Designed to collect participants' demographic and clinical characteristics.

Muscle Cramp Severity and Frequency Scale: This tool will assess the frequency and severity of muscle cramps. Developed based on a literature review, the scale records the date and frequency of cramps. Cramp episodes are defined according to the literature as involuntary leg movements lasting longer than one minute in hemodialysis patients. The number of episodes experienced during each dialysis session will be recorded.

Renal Function Tests: Parameters such as serum creatinine and urea levels will be evaluated.

Chronometer: A calibrated chronometer will be used to measure cramp duration, recorded in minutes.

Interventions Foot Massage Application: Participants will receive a 20-minute foot massage. The massage will be applied during dialysis treatment using techniques that support circulation to enhance tissue oxygenation and remove metabolic waste.

Foot Massage Protocol Before starting, the feet will be evaluated. Then, the feet will be cleaned with a wet compress and dried before proceeding with the massage. The total duration will be 20 minutes, with 10 minutes per foot. The massage will include five manipulation techniques: effleurage, petrissage, friction, percussion, and vibration, with only effleurage, petrissage, and friction used in this study.

Effleurage (Stroking): A light stroking movement over the skin. The massage starts and ends with effleurage, applying minimal pressure with the whole palm in a slow and steady motion using one or both hands. The fingers, except the thumbs, remain close together. Effleurage lasts approximately 2 minutes.

Petrissage (Kneading): The foot is kneaded by compressing and releasing it with both hands. This technique lasts around 3 minutes.

Friction: Circular and elliptical pressing and gliding movements are applied with the fingertips, from the sole to the dorsum of the foot, using varying pressures. This technique is performed for 5 minutes using the fingertips of the index or middle finger. The movement progresses towards the heart in small circular motions while applying adequate pressure.

Progressive Muscle Relaxation Exercises (PMRE): A 20-minute PMRE session will be conducted by the researcher. Participants will systematically tense and relax muscle groups throughout their bodies while undergoing dialysis treatment.

Progressive Muscle Relaxation Protocol

Before starting, participants will be given detailed information about the process. The exercises will focus on major muscle groups and follow these steps:

Foot Muscles: The foot muscles will be tensed for 5 seconds and then relaxed. Leg Muscles: The calf and thigh muscles will be stretched and relaxed in various positions.

Arm and Shoulder Muscles: The arms will be stretched forward and sideways, relaxing the muscles with active and passive relaxation movements.

Face and Neck Muscles: The forehead, jaw, and neck muscles will be tensed and then relaxed.

Duration and Repetitions: Each movement will involve 5-10 seconds of tension and 10-15 seconds of relaxation, with the entire protocol lasting approximately 20 minutes.

Completion: The session will conclude with deep breathing and relaxation exercises.

Both interventions will be applied twice a week for three weeks.

Control Group Participants in the control group will receive only routine hemodialysis treatment. They will not be exposed to any additional interventions during the data collection process.

Data Collection and Evaluation Study data will be collected at two time points: before the intervention (Day 1) and after the intervention (at the end of the 3rd week). The severity and frequency of muscle cramps will be assessed using the demographic information form and muscle cramp assessment scale. Blood tests will be conducted to measure serum creatinine and urea levels.

ELIGIBILITY:
Inclusion Criteria:

* Receiving Hemodialysis Treatment: Patients who have been undergoing regular hemodialysis treatment for at least six months.

History of Muscle Cramps: Patients who have experienced muscle cramps at least twice a week in the past month.

Age Range: Between 18 and 75 years old. Must be able to swallow tablets Cognitive and Physical Suitability: Having the cognitive and physical capacity to understand and perform massage and progressive muscle relaxation exercises.

Stable Cardiovascular Condition: No history of myocardial infarction or severe cardiovascular complications in the past three months.

Stable Medical Condition: No acute or severe medical conditions other than dialysis treatment.

Voluntary Participation: Signing the informed consent form after being fully informed about the study.

Exclusion Criteria:

Insulin dependent diabetes Thyroid disease Clinical diagnosis of Alzheimer's Disease

* Neuromuscular Disorders: Presence of conditions such as multiple sclerosis, Parkinson's disease, or peripheral neuropathy.

Severe Cardiovascular Diseases: History of myocardial infarction, congestive heart failure (NYHA class III-IV), or uncontrolled hypertension in the past three months.

Severe Orthopedic or Rheumatic Conditions: Severe osteoarthritis, rheumatoid arthritis, or other chronic musculoskeletal disorders.

Acute Infections or Inflammatory Conditions: Diagnosis of an active infection or inflammatory disease during the study period.

Mental or Psychiatric Disorders: Presence of severe cognitive impairment, dementia, or major depression/anxiety.

End-Stage Cancer Diagnosis: Undergoing active cancer treatment or having metastatic cancer.

Contraindications to Massage or Relaxation Exercises: Presence of skin infections, open wounds, or any medical condition preventing massage or exercise application.

Regular Use of Alternative Therapies: Engaging in regular massage therapy, yoga, or similar relaxation techniques within the past three months.

Pregnancy: Being pregnant or in the breastfeeding period. Inability to Comply with the Study: Difficulty in attending the study regularly or adhering to the assigned interventions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-05 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
pain report | 3 months
  pain measurement scale report

CONTACTS AND LOCATIONS:
Overall Officials: gürcan solmaz, Study Director — Istanbul University - Cerrahpasa

IPD SHARING:
Plan to Share IPD: No